CLINICAL TRIAL: NCT01687946
Title: Pilot Investigation on the Combined Use of Established Clinical Criteria and Systems Biology for Progressive Pulmonary Fibrosis
Brief Title: Explorative Study on the Molecular Pathology of Lung Fibrosis by Combination of Clinical Assessment and System Biology
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rolf Ziesche, Associated Professor of Medicine, Medical University of Vienna
Other Study IDs: RESOLVE - WP2; HEALTH-F4-2008-202047 (Other Grant/Funding Number: EC FP7 Health - Research Grant number HEALTH-F4-2008-202047)
Record Dates: First submitted 2012-08-23; First posted 2012-09-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Fibrosis
Keywords: Biology of Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Transbronchial biopsies and Video-assisted throracoscopic biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pulmonary fibrosis in aged individuals: Group A and B:
  Patients with UIP (histologically and/or radiologically proven) providing informed consent. According to functional and radiological assessment, the disease may be either limited (Group A) or advanced (Group B). The patients are usually older than 55 years.
- Pulmonary fibrosis and inflammation: Groups C and D:
  Patients with HP (histologically and radiologically proven) providing informed consent. According to functional and radiological assessment, the disease will be either acute or chronic. The patients will be significantly younger (mean > 10 years) than in groups A and B.
- Regular wound healing in lung: Patients receiving lung biopsy or bronchoscopy for reasons other that the study and volunteers providing informed consent. The group will consist of young (18-40 years) and old individuals (older than 55 years).

SUMMARY:
RESOLVE's objective is to identify and characterize validated molecular targets capable of shifting primary organ repair towards fibroproliferative wound healing.

Work package 2 (WP2) of RESOLVE includes the clinical study protocols within the RESOLVE system evaluating different forms of pulmonary repair in humans ranging from normal repair over mainly inflammatory to predominantly fibroproliferative repair.

Hypothesis

Fibrosis of the lung is an aberrant and intensified form of wound healing. It is the result of an unresolved disturbance of both initiation and control of repair which is partly age-related. As a result of the relentlessly activated wound healing reaction, mechanisms of inflammation largely representing the condition of chronic inflammation within the peripheral bronchial tree will aggravate this abnormal form of repair.

A systematic comparison of the molecular pathology of fibrotic repair representing

* Varying intensity of fibrosis related to the pathology of usual interstitial pneumonia (UIP),
* Varying inflammatory mechanisms (UIP vs. Hypersensitivity pneumonitis [HP], acute and chronic), and
* Varying stages of age (Normal pulmonary repair in young and old individuals vs. acute/chronic HP vs. UIP) will be able to
* identify molecules capable of shifting regular repair towards fibroproliferative repair and
* elucidate their interrelationship with other molecules forming coordinated yet misdirected metabolic responses characteristic for fibroproliferative repair.

DETAILED DESCRIPTION:
Background

After reaching adulthood, the organs of the human body preserve their shape and function over a long period, making directed repair one of the most important mechanisms throughout lifetime. Regular wound healing after an injury consists of a well-ordered sequence of overlapping phases: inflammation, formation of supportive new tissue, re-epithelization and final regeneration of epithelial and endothelial lining cells, and essentially repeats the complex process of organ development. In young adults, damage to an organ is frequently answered by fully regenerative wound healing repeating mechanisms of embryonic organ growth called "primary" wound healing. Repeated damage in younger individuals may cause "secondary" wound healing in form of scar formation serving as a rescue program to maintain surface integrity once epithelial and/or endothelial reorganization has failed.

Organ failure in the ageing organism, however, is different and essentially represents the loss of its capacity to achieve an orderly reactivation of organ development. This different quality of wound healing consists of a combination of chronic inflammation and fibroproliferative, non-regenerative repair. Its pathology refers to a large group of diseases involving every organ of the human body.

In the lung, its most prominent form is characterized by a well-defined histopathology named usual interstitial pneumonia (UIP). Unfortunately, this histopathology, while identifying a particularly aggressive phenotype of the fibroproliferative repair response itself, does not allow for an unambiguous clinical diagnosis, as the UIP "pattern" may be found in different fibrotic diseases of the lung, such as hypersensitivity pneumonitis (HP), especially in its chronic form.

In addition, various mechanisms of inflammation which are partly related to the wound healing response itself, may profoundly intensify the aberrant wound healing response. As a result, the mechanisms leading to this condition and maintaining its characteristic clinical appearance are unknown.

The current investigation belongs to the work package 2 of the RESOLVE study system (FP7-HEALTH-F4-2008 Contract no. 202047) which contains the clinical study protocol evaluating different forms of fibrotic repair in the human lung. RESOLVE's main objective is to identify and characterize clinically validated molecular targets capable of shifting primary organ repair towards fibroproliferative wound healing. In this pilot study, different forms of repair of the lung will be prospectively analyzed by means of a concomitant clinical and biological analysis guided by evaluated functional and radiological measures of clinical development. The assessments will be made at the beginning of the study period (visit 1), after three months of prospective observation (visit 2), and after 12 months (end of study) allowing for a clinically relevant correlation of all biological data obtained.

Three general conditions of repair will be chosen for systematic biological analysis as a result of their clinical diagnosis (histopathology, radiology) and their association with age:

* Usual interstitial pneumonia (UIP) occurring almost exclusively at an age of 55-80 years,
* Hypersensitivity Pneumonitis (HP), both acute and chronic, occurring at an age of 20-55 years, and
* Normal repair in young (18-40 years) and old (older than 55 years) individuals.

Methods

After securing the diagnosis (see below: inclusion/exclusion criteria) and following informed consent during the screening visit, patients lacking any previous immunosuppressive treatment (therapy-naïve patients) will receive an immunosuppressive therapy with prednisolone (daily dose of 1 mg/kg BW) for at least three months in order to exclude pathologies dominated by mechanisms of inflammation. During the screening visit, the results of the histopathological analysis will be secured, and the clinical and functional history of the disease recorded. This will include previous medication, the results of previous pulmonary function tests (PFT) as well as the results of radiological analysis (computed tomography including HR-CT) and lab testing (excluding collagen vascular disease and securing HP serology).

Three months after the screening visit, at visit 1, the functional and radiological stage of the pulmonary fibrosis will be assessed again, and the patients will be finally enrolled into the study. In accordance with the findings obtained at the screening visit, and due to the functional and radiological results obtained at visit 1, the patients will be stratified into the following investigational groups:

Group A:

(Limited UIP) Patients with proven UIP and functionally and radiologically less advanced pulmonary fibrosis (n=12) as defined by histopathology (assessment by two independent and experienced pathologists not involved in the study) and/or radiology (computed tomography [CT] scans incl. high-resolution CT, independently assessed by an experienced radiologist not involved in the study) and pulmonary function tests (PFT). PFT will consist of spirometry, measurement with bodyplethysmograph, single-breath measurement of carbon monoxide diffusion capacity and full cardiopulmonary exercise testing including assessment of pulmonary ventilation and gas exchange at rest and on exertion;

Group B:

(Advanced UIP) Patients with proven UIP (n=12) in a significantly more advanced stage of the disease as determined by PFT (FVC at least 10 percent and DLCO at least 15 percent lower than in group A) and CT scan;

Group C:

(Chronic fibrosing Hypersensitivity Pneumonitis, HP) Patients with chronic fibrosing HP (n=12) diagnosed by histopathology, radiology and lab testing;

Group D:

(Acute HP) Patients with acute HP (n=9) diagnosed by histopathology, radiology and lab testing (Group D: acute HP);

Group E:

Regular Pulmonary Repair 9 young (18-40 years of age) without any clinically evident pathology and 9 old volunteers (55-80 years of age) without pulmonary fibrosis will serve as controls.

All patients with UIP and HP will be followed during for a study period of 12 months. The study period starts with visit 1. In addition to visit 1, two additional visits will be performed after 3 months (visit 2, functional assessment) and after 12 months (visit 3, end of study).

At all three visits, the following investigations will be performed:

* Clinical examination
* ECG
* PFT
* Cardiopulmonary exercise test
* Blood drawing
* CT scan
* Bronchoscopy with removal of 5 transbronchial biopsies for biological assessment from areas suggesting maximum disease activity in the CT scan will only be performed at visits 1 and 3.

Relevant inclusion criteria applying to Group A (limited UIP):

* Informed consent
* Histologic proof of lesions consistent with UIP in surgical lung biopsies and/or
* Radiological signs suggestive of UIP
* No signs of widespread ground-glass opacities in CT scans
* No symptoms suggestive of chronic bronchitis/bronchiolitis, such as coughing and signs of bronchial obstruction or hyperinflation
* Difference of forced expiratory vital capacity (FVC) values ≤ 10% predicted to normal
* Difference of carbon monoxide diffusion capacity (DLCO) at rest of ≤ 15% predicted to normal
* Previous or current treatment with immunosuppressive drugs

Relevant inclusion criteria applying to Group B (advanced UIP) (other than Group A):

* Signs of widespread ground glass opacities in CT scans
* Symptoms suggestive of chronic bronchitis, such as coughing and signs of bronchial obstruction or hyperinflation, may be present
* Forced expiratory vital capacity (FVC) values in difference > 10% predicted to normal
* Reduction of carbon monoxide diffusion capacity (DLCO) at rest of < 15% predicted

Relevant inclusion criteria applying to Group C:

* Informed consent
* Histologic and/or cytologic proof of lesions consistent with chronic HP in transbronchial and/or surgical lung biopsies, transbronchial biopsies or bronchoalveolar lavage (BAL) samples
* Radiological signs suggestive of chronic HP
* Signs of widespread ground glass opacities in CT scans
* Symptoms suggestive of active bronchitis/bronchiolitis, such as coughing and signs of bronchial obstruction or hyperinflation, may be present
* Serological proof of hypersensitivity, if possible
* Forced expiratory vital capacity (FVC) values in difference ≥ 10% predicted to normal
* Reduction of carbon monoxide diffusion capacity (DLCO) at rest of ≥ 15% predicted
* Previous or current treatment with immunosuppressive drugs

Relevant inclusion criteria applying to Group D (other than Group C):

* Informed consent
* Histologic and/or cytological proof of lesions consistent with acute HP in transbronchial and biopsies and/or bronchoalveolar lavage (BAL) samples
* Radiological signs suggestive of acute HP

General exclusion criteria

* Functionally significant cardiovascular morbidity
* Respiratory insufficiency (PaO2 < 55 mmHg; PaCO2 > 50 mmHg)
* Significant pulmonary hypertension
* Significant pulmonary emphysema
* Non-functional contralateral lung
* Cancer
* Significant coronary heart disease
* Coagulation dysfunction
* Pregnancy, or planning pregnancy during the trial or within three month period thereafter
* Known drug or alcohol abuse within 3 years of screening
* Presumed non-compliance
* Known legal incapacity or limited legal capacity at screening

Biopsies

The lung specimens for biological analysis will be derived from both diagnostic surgical lung biopsies and transbronchial lung biopsies taken during the bronchoscopies performed at visit 1 and 3. In total, five transbronchial biopsies will be taken at each visit for biological analysis. All transbronchial lung specimens will be removed under radiologic control from peripheral lung areas previously specified in accordance with the latest CT scan. The biopsies taken at visit 3 will be performed in the same lung segment as those taken at visit 1.

Except for the results of the latest CT scan, the investigator performing the bronchoscopy will be blinded for all clinical results obtained during the visits.

Molecular Biology Assessment

Biological analysis will be independently performed. All investigators involved in biological analysis will be blinded for diagnosis and clinical course of the patients and volunteers. The participants will be solely identifiable by their study identification number (ID). The study samples will be numbered according to patient ID and sample description provided by the LIMS. Biologic assessment will include measurement of whole genome transcriptomics, protein analysis by mass spectrometry and EIA, analysis of DNA methylation status, and microRNA analysis. The measurements will be based on lung specimens derived from diagnostic surgical lung biopsies, if possible, and/or from transbronchial biopsies (TbX) taken during a bronchoscopy at visit 1 and 3 of the study (month 0 and month 12). In addition, BAL fluid will be stored and used for detection of proteins and lipids. Materials for DNA methylation analysis will be obtained from both lung tissue and whole blood samples.

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Histological and radiological proof of UIP or HP

Exclusion criteria

* Functionally significant cardiovascular morbidity
* Respiratory insufficiency (PaO2 < 55 mmHg; PaCO2 > 50 mmHg)
* Significant pulmonary hypertension
* Significant pulmonary emphysema
* Non-functional contralateral lung
* Cancer
* Significant coronary heart disease
* Coagulation dysfunction
* Pregnancy, or planning pregnancy during the trial or within three month period thereafter
* Known drug or alcohol abuse within 3 years of screening
* Presumed non-compliance
* Known legal incapacity or limited legal capacity at screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants are chosen from patients lists of participating center.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Analysis of lung biopsies by system biology techniques. | Two measurements within 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Lutz H Block, MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No